CLINICAL TRIAL: NCT02759393
Title: Comparing Dexlansoprazole With Double-dose Lansoprazole to Achieve Sustained Symptomatic Response in Overweight and Obesity Patients With Reflux Esophagitis in Los Angeles Grades A & B
Brief Title: Treatment Effect Between Dexlansoprazole and Double-dose Lansoprazole in Obesity Patients With Reflux Esophagitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHW104-TDU-B-2111-113002
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEX group (Experimental): receiving 8-week dexlansoprazole 60 mg per day
  Interventions: Drug: Dexlansoprazole
- Double-dose PPI group (Active Comparator): receiving 8-week lansoprazole 30 mg twice daily
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — receiving 8-week PPI
  Arms: DEX group
Drug: Lansoprazole — receiving 8-week PPI
  Arms: Double-dose PPI group

SUMMARY:
The purpose of this study is to investigate whether dexlansoprazole can be as effective as double dose PPI to achieve SSR in high BMI cases with reflux esophagitis in Los Angeles grades A & B.

DETAILED DESCRIPTION:
This study is conducted in National Cheng Kung University Hospital, a tertiary health care center in Tainan, Taiwan. All participants give written informed consent before enrollment. After panendoscopy to confirm enrollment eligibility and reflux esophagitis in Los Angeles A or B, all patients are evenly randomized into a DEX group (receiving 8-week dexlansoprazole 60 mg per day) or double-dose PPI group (receiving 8-week lansoprazole 30 mg twice daily). The enrolled patients are randomized by two series of sealed envelopes containing a prescheduled group code; one series for the overweight patients and the other for the obese patients. In each series of the sealed envelopes, the number of the group code will be equal within every 10 sealed envelopes.

In each patient, the demographic factors and the genotype of S-mephenytoin 4'-hydroxylase (CYP2C19) will be checked and defined as poor metabolizer (PM), homologous (HomoEM) or heterologous extensive metabolizer (HeteroEM). Each patient is treated continuously with dexlansoprazole 60 mg per day or lansoprazole 30 mg twice daily for eight weeks. During this 8-week study period, each patient is requested to record their daily clinical symptoms of reflux esophagitis on a special sheet, including the severity of acid regurgitation (AR, score 0: free from symptoms; score 1: attack episodes < 5 times per day; score 2: 6-10 times per day; score 3: more than 10 episodes per day), heartburn (HB, score 0: absence of symptoms; score 1: tolerable events not interfering with daily work; score 2: intolerable events interfering with daily work, but not needing medication to relieve the symptoms; score 3: complaints interfering with the completion of daily work, or causing the patient to wake up during the night with cough, or combined with any other non-specific complaints). The patients are scheduled to return to clinics for drug refills, and to hand back daily symptom records at the end of the fourth and eighth week of treatment.

The cumulative proportions of patients with sustained symptomatic response (SSR), defined as free from acid regurgitation and heartburn for the last seven days, are recorded during the 8-week study period for each study group. All of the patients starting the treatment are included for the intention-to-treat (ITT) analysis of the rate of SSR. If patients have obvious symptoms despite continuous PPI usage and have an unscheduled visit to load up on additional PPIs during the study, the case is then dropped from the per-protocol (PP) analysis. In addition, patients lost to follow-up are excluded from the PP analysis to determine the rate of SSR. Besides comparing the difference of the rate of SSR between the two study groups, the study also determined whether patients with different CYP2C19 genotypes have differences in the cumulative rates of SSR after therapy between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants included patients ≥20 years with either overweight (BMI of 25-30 kg/m2) or obese (BMI > 30 kg/m2), who had undergone panendoscopy due to typical clinical symptoms of either acid regurgitation, heartburn sensation, or both. By the results of panendoscopy, patients with the severity of grade A or B esophageal reflux, according to the Los Angeles classification, are enrolled.

Exclusion Criteria:

* Patients are excluded if they have taken antisecretory agents, including histamine-2 receptor antagonist and PPI, within two weeks prior to the panendoscopy. The following conditions are also excluded: the presence of peptic ulcers, pregnancy, major medical problems (including hypertension, liver cirrhosis, COPD, asthma, renal failure and congestive heart failure), or previous gastric surgery. Patients who have an allergy history to dexlansoprazole or lansoprazole are also excluded.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the rate of sustained symptomatic response (SSR) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Shyang Sheu, MD, Study Director — National Cheng-Kung University Hospital

REFERENCES:
- [Background] Jacobson BC, Somers SC, Fuchs CS, Kelly CP, Camargo CA Jr. Body-mass index and symptoms of gastroesophageal reflux in women. N Engl J Med. 2006 Jun 1;354(22):2340-8. doi: 10.1056/NEJMoa054391. PMID 16738270
- [Background] Hampel H, Abraham NS, El-Serag HB. Meta-analysis: obesity and the risk for gastroesophageal reflux disease and its complications. Ann Intern Med. 2005 Aug 2;143(3):199-211. doi: 10.7326/0003-4819-143-3-200508020-00006. PMID 16061918
- [Background] Sheu BS, Cheng HC, Chang WL, Chen WY, Kao AW. The impact of body mass index on the application of on-demand therapy for Los Angeles grades A and B reflux esophagitis. Am J Gastroenterol. 2007 Nov;102(11):2387-94. doi: 10.1111/j.1572-0241.2007.01468.x. PMID 17850409
- [Background] Chen WY, Chang WL, Tsai YC, Cheng HC, Lu CC, Sheu BS. Double-dosed pantoprazole accelerates the sustained symptomatic response in overweight and obese patients with reflux esophagitis in Los Angeles grades A and B. Am J Gastroenterol. 2010 May;105(5):1046-52. doi: 10.1038/ajg.2009.632. Epub 2009 Nov 10. PMID 19904250
- [Background] Peura DA, Pilmer B, Hunt B, Mody R, Perez MC. Distinguishing the impact of dexlansoprazole on heartburn vs. regurgitation in patients with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2013 Nov;38(10):1303-11. doi: 10.1111/apt.12504. Epub 2013 Sep 30. PMID 24118079
- [Background] Peura DA, Pilmer B, Hunt B, Mody R, Perez MC. The effects of increasing body mass index on heartburn severity, frequency and response to treatment with dexlansoprazole or lansoprazole. Aliment Pharmacol Ther. 2013 Apr;37(8):810-8. doi: 10.1111/apt.12270. Epub 2013 Mar 4. PMID 23451835
- [Background] de Morais SM, Wilkinson GR, Blaisdell J, Nakamura K, Meyer UA, Goldstein JA. The major genetic defect responsible for the polymorphism of S-mephenytoin metabolism in humans. J Biol Chem. 1994 Jun 3;269(22):15419-22. PMID 8195181
- [Background] Sheu BS, Kao AW, Cheng HC, Hunag SF, Chen TW, Lu CC, Wu JJ. Esomeprazole 40 mg twice daily in triple therapy and the efficacy of Helicobacter pylori eradication related to CYP2C19 metabolism. Aliment Pharmacol Ther. 2005 Feb 1;21(3):283-8. doi: 10.1111/j.1365-2036.2005.02281.x. PMID 15691303